CLINICAL TRIAL: NCT03813134
Title: EURO SHOCK Testing the Value of Novel Strategy and Its Cost Efficacy in Order to Improve the Poor Outcomes in Cardiogenic Shock
Brief Title: Testing the Value of Novel Strategy and Its Cost Efficacy in Order to Improve the Poor Outcomes in Cardiogenic Shock
Acronym: EUROSHOCK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leicester (Other)
Collaborators: European Commission (Other); University of Glasgow (Other); KU Leuven (Other); University of East Anglia (Other); Deutsches Herzzentrum Muenchen (Other); A.O. Ospedale Papa Giovanni XXIII (Other); Chalice Medical Ltd (Unknown); Ludwig-Maximilians - University of Munich (Other); University of Tromso (Other); Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other); Paula Stradina Liniska Universitates (Unknown); Accelopment AG (Other); Universiteit Antwerpen (Other); European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0658
Record Dates: First submitted 2018-12-19; First posted 2019-01-23 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Cardiogenic Shock
Keywords: Cardiogenic Shock; Acute Myocardial Infarction; Acute Coronary Syndrome
MeSH Terms: conditions — Shock, Cardiogenic; Acute Coronary Syndrome | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: Prospective, open, multicentre, randomised strategy trial in Cardiogenic Shock (CGS)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate PCI with medical therapy (Active Comparator): Group 1 will receive immediate revascularisation with Percutaneous Coronary Intervention (PCI) to the culpirit lesion only) + standard care (pharmacological support titrated to attain SBP >90mmHg).
  No mechanical support device allowed.
  Interventions: Procedure: Percutaneous coronary intervention (PCI); Other: Pharmacological Support
- Immediate PCI with early VA-ECMO (Experimental): Group 2 will receive immediate PCI plus standard pharmacological support with early peripheral veno-arterial ECMO.
  Interventions: Procedure: Percutaneous coronary intervention (PCI); Other: Pharmacological Support; Device: VA-ECMO

INTERVENTIONS:
Procedure: Percutaneous coronary intervention (PCI) — Primary PCI or early/immediate PCI for NSTEMI will be undertaken according to recommended Guideline standards of care. This will include appropriate pre-loading with dual anti-platelet therapy, a preferred radial approach, intra-procedural anti-coagulation (with measure of ACT if considered appropriate every 30 minutes) and the use of drug eluting stents. Treatment will be delivered essentially to the culprit vessel only. A successful procedure will be one considered to have achieved TIMI 2-3 flow and residual stenosis < 50%. PCI failure will not be an exclusion itself from the trial.
Other: Pharmacological Support — Use of pharmacological agents (Norepinephrine, Dobutamine, Levosimendan) according to ESC Guidelines to maintain mean arterial pressure >75 mmHg in accordance with recognised standards of care. Changes in pharmacotherapy will NOT be regarded as escalation therapy. However the number of and dose of inotropes will be documented in the CRF.
Device: VA-ECMO — Following PCI of the culprit lesion, patients will have ECMO initiated as soon as echocardiography (to exclude mechanical causes) has been completed, once they have been assessed as having failed to improve (with the aim to start ECMO as early as possible from 30 mins after completed P-PCI procedure ad fully established within 6 hours after randomisation).
  Peripheral Veno-arterial ECMO will be employed with a flow rate according to individual patient needs. Other methods of LV unloading, distal limb perfusion, maintenance of ejection/aortic valve opening and anti-coagulation will be instituted as per sites' usual care.
  A minimum 24 hours be allocated to the randomised therapy in order that strategy failure is demonstrated but this will be at the physicians' discretion.
  Other Names: Veno-Arterial Extra Corporeal Membrane Oxygenation.
  Arms: Immediate PCI with early VA-ECMO

SUMMARY:
Cardiogenic shock (CGS) affects up to 10% of patients suffering acute coronary syndrome. It has a 30 day mortality of 45-50%. No pharmacological nor intervention/device trials have had any impact on this mortality in the last 20 years.

The EURO SHOCK Trial (supported by the European Union Horizons 2020 programme) will randomise 428 patients with CGS following acute coronary syndrome from 44 EU centres to early intervention with Extra Corporeal Membrane Oxygenation (ECMO) therapy or to standard treatment (with no ECMO). This intervention is a high cost specialist centre procedure that warrants further investigation including economic appraisal. Multiple mechanistic and hypothesis generating sub-studies will be undertaken.

DETAILED DESCRIPTION:
The EURO SHOCK trial tests the novel use of early deployment of mechanical support device in Cardiogenic Shock (CGS) in a randomised, strategy trial, with evidence of benefit or otherwise measured by recording hard clinical end-point outcomes.

Extra Corporeal Membrane Oxygenation (ECMO) is already used in CGS. This is therefore not a novel therapy. It is the use of ECMO early in the development of CGS that is the novel aspect of this project. The Investigators will test whether a strategy of very early ECMO can ameliorate the rapid decline that many CGS patients suffer. The value of deploying a clinically used and approved device prospectively and early in the natural history of CGS compared to standard practice has not been tested before and will be the basis of the EURO SHOCK project.

This trial itself will be a prospective randomized, open label, design study that will compare two groups of patients: Both will receive appropriate percutaneous coronary intervention (PCI) as is current practice as they arrive at the hospital.

1. Group 1 will receive immediate PCI + standard care (pharmacological support).
2. Group 2 will receive immediate PCI plus support with early peripheral veno-arterial ECMO + standard care (pharmacological support).

The Investigators will also compare the cost-effectiveness of early VA-ECMO, as compared to current standard of care. EURO SHOCK will also evaluate novel CMR protocols in these unwell patients, and also whether systems of urgent flagged transfer of the unwell patient is practical and beneficial. The Investigators will determine whether there are biological and ECG markers that predict worse patient outcomes, which could thus help select most appropriate patients for expedited treatments (the patient is only transferred if needed).

Although at the centre of the project there is a randomised trial, other important objectives will therefore be delivered.

The research study will additionally focus, through a-priori, post-hoc analyses, on higher risk and vulnerable sub groups such as the elderly (>75 years) and females, the importance of site of infarct and on those with multi-morbidities such as diabetes. These post-hoc data will be published separately.

The trial will include patients with out of hospital cardiac arrest (OHCA) who have documented return of spontaneous circulation (ROSC) but with certain caveats (see exclusion criteria).

The primary outcome is the all-cause mortality at 30 days following admission with acute coronary syndrome with cardiogenic shock. Key secondary outcomes will include all- cause mortality or admission with heart failure at 12 months, all-cause mortality at 12 months and admission to hospital with heart failure at 12 months.

A cornerstone of this research programme will be to determine the cost-efficacy of ECMO in this setting. Cost benefit will be measured both immediately and in the longer term testing for example any impact of need for heart failure therapies. This will be undertaken with evaluations of the cost-effectiveness of the device and evaluation of quality of life using the EuroQuol-5D-5L and the Minnesota Living with Heart Failure Questionnaire.

The EUROSHOCK trial will also include the following sub-studies:

1. Cardiovascular MRI: Cardio-Renal Imaging Sub-study using novel shortened, non-breath-holding protocols.
2. Platelet Function Sub-study designed to access the impact of novel ECMO coatings on platelet activation.

The programme will be developed and run through a carefully thought through management structure comprising 8 separate but interlinked work programmes (each targeted at one aspect of the project and headed by an experienced clinical trialist or trial manager) and involve the dissemination of results through a designated dissemination work package. Attention to translating the results to subsequent on-the-ground patient care will be an important aim for the management and dissemination team, and will involve patient support groups, professional societies and information delivered directly to the medical and non- medical staff caring for CGS patients.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to provide informed consent/assent.
2. Presentation CGS within 24 hours of onset of Acute Coronary Syndrome (ACS) symptoms.
3. CGS can only be secondary to ACS (Type 1 MI STEMI or N-STEMI) or secondary to ACS following previous recent PCI (acute/sub-acute stent thrombosis ARC)
4. PCI has been attempted.
5. Persistence of CGS 30 minutes after successful or unsuccessful revascularisation of culprit coronary artery to allow for echocardiography and clinical assessment.

   CGS will be defined by the following 2 criteria:

   • Systolic blood pressure <90 mmHg for at least 30 minutes, or a requirement for a continuous infusion of vasopressor or inotropic therapy to maintain systolic blood pressure > 90 mmHg.

   Clinical signs of pulmonary congestion, plus signs of impaired organ perfusion with at least one of the following manifestations:
   * altered mental status.
   * cold and clammy skin and limbs.
   * oliguria with a urine output of less than 30 ml per hour.
   * elevated arterial lactate level of >2.0 mmol per litre.
6. Provision of informed assent followed by patient consent; [or relative or physician consent if the patient is unable to consent].

Exclusion Criteria:

1. Unwilling to provide informed assent/consent.
2. Echocardiographic evidence) of mechanical cause for CGS: eg ventricular septal defect, LV-free wall rupture, ischaemic mitral regurgitation (recorded within 30 mins of end of PCI procedure).
3. Age <18 and>90 years.
4. Deemed appropriately frail (≥ 5 Canadian frailty score)
5. Shock from another cause (sepsis, haemorrhagic/hypovolaemic shock, anaphylaxis, myocarditis etc.).
6. Significant systemic illness
7. Known dementia of any severity.
8. Comorbidity with life expectancy <12 months.
9. Severe peripheral vascular disease (precluding access making ECMO contra- indicated).
10. Severe allergy or intolerance to pharmacological or antithrombotic anti-platelet agents.
11. Out-of-hospital cardiac arrest (OHCA) under any of the following circumstances:-

    * without return of spontaneous circulation (ongoing resuscitation effort).
    * without pH or >7 without bystander CPR within 10 minutes of collapse.
12. Involved in another randomised research trial within the last 12 months.
13. Arterial lactate level of <2.0 mmol per litre.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Estimated)
Dates: Start 2019-10-11 (Actual); Primary Completion 2023-03-03 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality at 30 days | at 30 days
  Death from any cause

SECONDARY OUTCOMES:
All-cause mortality or admission for heart failure at 12 months | at 12 months
  Death from any cause, or admission to hospital for heart failure with typical symptoms (e.g. breathlessness, ankle swelling and fatigue) that may be accompanied by signs (e.g. elevated jugular venous pressure, pulmonary crackles and peripheral oedema) caused by a structural and/or functional cardiac abnormality, resulting in a reduced cardiac output and/or elevated intracardiac pressures at rest or during stress.
All-cause mortality at 12 months | at 12 months
  Death from any cause
Admission for heart failure at 12 months | at 12 months
  Admission to hospital with clinical syndrome of heart failure, defined as per the ESC guidelines as typical symptoms (e.g. breathlessness, ankle swelling and fatigue) that may be accompanied by signs (e.g. elevated jugular venous pressure, pulmonary crackles and peripheral oedema) caused by a structural and/or functional cardiac abnormality, resulting in a reduced cardiac output and/or elevated intracardiac pressures at rest or during stress.

OTHER OUTCOMES:
All-cause mortality | From date of index hospital admission to date of discharge from hospital, assessed up to 12 months.
  Death from any cause
Cardiovascular mortality | From date of index hospital admission to date of discharge from hospital, assessed up to 12 months.
  Death due to cardiovascular causes, including myocardial infarction, heart failure, cardiac arrhythmias, stroke, and sudden death suspected from cardiac aetiology.
Stroke. | From date of index hospital admission to date of discharge from hospital, assessed up to 12 months
  Acute neurological deficit lasting longer than 24 hours. The type of stroke will be categorised as: 1) Primary Haemorrhagic: either intracranial haemorrhage or subdural haematoma. 2)non-hemorrhagic cerebral infarction. 3)non-hemorrhagic cerebral infarction with haemorrhagic conversion. 4)Uncertain (any stroke without brain imaging [CT or MRI] or autopsy definition of type, or if tests are inconclusive).
Recurrent Myocardial Infarction | From date of index hospital admission to date of discharge from hospital, assessed up to 12 months.
  Defined as the presence of ischaemic symptoms of angina-type pain lasting longer than 20mins, its evidence of either ST-segment elevation/new Left Bundle Branch Block on ECG, or evidence of new Troponin elevation by greater than 20% of the last non-normalised reading, or angiographic evidence of re-occlusion of a previously opened artery or graft.
Bleeding (BARC Type 3-5) | From date of index hospital admission to date of discharge from hospital, assessed up to 12 months.
  Evidence of Bleeding as per the Bleeding Academic Research Consortium classification Type 3, Type 4 or Type 5.
Escalation to other (non-ECMO) support device for refractory shock | From date of index hospital admission to date of discharge from hospital, assessed up to 12 months.
  The use of either Impella or Tandem-Heart or LVAD support devices in patients with persistent cardiogenic shock despite revascularisation and uptitation of pharmacological support. Use of ECMO or non ECMO MSD in standard care group or to non ECMO device in intervention (ECMO) group will be regarded as a protocol violation and managed statistically as such in the final analysis.
Any vascular complications | From date of index hospital admission to date of discharge from hospital, assessed up to 12 months.
  Complications affecting the peripheral vasculature, defined by the Valve Academic Research Consortium (VARC)-2 classifications.
Acute Kidney Injury according to the modified RIFLE classification | From date of index hospital admission to date of discharge from hospital, assessed up to 12 months.
  Evidence of Acute Kidney Injury according to the RIFLE (Risk, Injury, Failure, Loss and End-stage kidney disease) classification stage 1 - 3.
MACCE (Major Adverse Cardiovascular and Cerebrovascular Events) | at 12 months
  combined endpoint of all-cause mortality, repeat MI, stroke and re-hospitalization for heart failure.
Cardiovascular mortality | at 12 months
  Death due to cardiovascular causes, including myocardial infarction, heart failure, cardiac arrhythmias, stroke, and sudden death from cardiac aetiology.
Recurrent Myocardial Infarction | at 12 months
  Defined as the presence of ischaemic symptoms of angina lasting longer than 20mins, its evidence of either ST-segment elevation/new Left Bundle Branch Block on ECG, or evidence of new Troponin elevation by greater than 20% of the last non-normalised reading, or angiographic evidence of re-occlusion of a previously opened artery or graft.
Stroke | at 12 months
  Acute neurological deficit lasting longer than 24 hours. The type of stroke will be categorised as: 1) Primary Haemorrhagic: either intracranial haemorrhage or subdural haematoma. 2)non-hemorrhagic cerebral infarction. 3)non-hemorrhagic cerebral infarction with haemorrhagic conversion. 4)Uncertain (any stroke without brain imaging [CT or MRI] or autopsy definition of type, or if tests are inconclusive).
Need for unplanned (Ischaemia-Driven) repeat revascularization (PCI and/or CABG) after index procedure [staged procedures excluded] | at 12 months
  REvascularisation procedure (either PCI or CABG) undertaken after index procedure in the context of ischaemic symptoms and evidence of myocardial ischaemia (ECG, stress perfusion scan, acute myocardial infarction) either to the culprit or non-culprit lesion. Planned elective staged procedures to the non-culprit lesion will not be included.
Failure of discharge from primary admission as measured at 30 days | at 30 days
  Patient remains an in-patient in hospital for on-going medical care following the index admission with acute coronary syndrome complicated by cardiogenic shock.
Bleeding (BARC Type 3-5) | at 12 months
  Evidence of Bleeding as per the Bleeding Academic Research Consortium classification Type 3, Type 4 or Type 5.
Infarct size on Cardiac Magnetic Resonance Imaging | From date of index hospital admission to date of discharge from hospital, assessed up to 12 months.
  The size of myocardial infarction, quantified as the percentage of myocaridum demonstrating late gadolinium enhancement consistent with acute myocardial injury.
Cost effectiveness | at 12 months
  The cost effectiveness of using early ECMO in patients with cardiogenic shock complicating acute myocardial infarction will be assessed using the Incremental Cost Effectiveness Ratio (ICER)
Quality of Life as assessed using the EuroQuol-5D-5L (measured at discharge, 6 and 12 months) | on day of discharge from hospital following index admission, at 6 months and at 12 months
  Assess the participants' general health status and self-reported quality of life using the EQ5D questionnaire. This is a 5 level EQ-5D standardised measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal.
  The EuroQuol (EQ)-5D-5L questionnaire assesses quality of life in study participants according to 5 domains (mobility, self care, usual activities, pain/discomfort, anxiety/depression) each scored according to a scale of 1 (no problems) to 5 (indicating extreme problems) and generating a 5-digit code corresponding to quality of life. This will be used at discharge, 6 months and 12 months, and the within-subject change in EQ-5D-5L scores will be measured for this secondary outcome.
Quality of Life assessed using the Minnesota Living with heart failure questionnaire (measured at discharge, 6 and12 months) | on day of discharge from hospital following index admission, at 6 months and at 12 months
  This is a standardised measure of quality of life for patients living with heart failure. The questionnaire includes 21 physical, emotional and socio-economic ways in which heart failure can adversely affect the patients life, each domain is scored from 0 to 5 indicating how much heart failure has prevented the patient from living how he or she wanted to live over the preceding 4 weeks. This will be assessed for each patient at time of discharge, at 6-months and again at 12 months. The within-subject change in the MLFHQ questionnaire will be measured for each group.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony H Gershlick, Principal Investigator — University of Leicester
Locations (47):
- Medical University of Vienna, Vienna, Vienna, Austria
- Belgium (10):
  - Algemeen Stedelijk Ziekenhuis Aalst, Aalst
  - Onze Lieve Vrouw Hospital Aalst, Aalst
  - University Hospital Antwerpen, Antwerp
  - ZNA Middelheim, Antwerp
  - Imelda Hospital Bonheiden, Bonheiden
  - AZ Monica, Deurne
  - AZ Gent, Ghent
  - Jessa Ziekenhuis Hasselt, Hasselt
  - Katholieke Universiteit Leuven, Leuven
  - AZ Turnhout, Turnhout
- Germany (10):
  - Universitäts-Herzzentrum Freiburg-Bad Krozingen, Bad Krozingen
  - Segeberger Kliniken GmbH, Bad Segeberg
  - Herz-Zentrum Bodensee, Konstanz
  - Klinikum Rechts Der Isar, Munich
  - Klinikum Campus Innenstadt, München
  - Deutsches Herzzentrum München, München
  - Barmherzige Brüder gemeinnützige Krankenhaus GmbH, München
  - Klinik Augustinum, München
  - Ludwig-Maximilians-Universität München, München
  - Uniklinikum Tübingen, Tübingen
- Italy (5):
  - Azienda Ospedalierea Papa Giovanni XXIII, Bergamo
  - University Hospital of Bologna Policlinico S. Orsola - Malpighi, Bologna
  - Azienda Universitaria Ospedaliera Careggi, Firenze, Florence
  - Università degli Studi di Padova, Padua
  - Ospedale San Giovanni Bosco di Torino, Torino
- Paula Stradina Liniska Universitates Slimnica AS, Riga, Latvia
- Norway (4):
  - The Nordland Hospital, Bodø
  - The Finnmark Hospital, Hammerfest
  - The Helgeland Hospital, Mo i Rana
  - Universitetet i Tromsoe, Tromsø
- Spain (5):
  - Hospital Germans Trias I Pujol, Badalona
  - Hospital Vall d'Hebron, Barcelona
  - Consorci Institut D'Investicacions Biomediques August Pi i Sunyer / Hospital Clinic de Barcelona, Barcelona
  - Hospital de Sant Pau, Barcelona
  - Hospital de Bellvitge, Barcelona
- United Kingdom (11):
  - University Hospital Leicester, Leicester, East Midlands
  - Hairmyres Hospital, Airdrie, Lanarkshire
  - University of Leicester, Leicester, Leicestershire
  - Newcastle Freeman Hospital, Newcastle, Newcastle Upon Tyne
  - University of Glasgow, Glasgow, Scotland
  - Papworth Hospital, Cambridge
  - Golden Jubilee National Hospital, Glasgow
  - St Barts and the London Hospital, London
  - Kings College Hospital, London
  - Harefield and Brompton London, London
  - Guys and St Thomas NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No